CLINICAL TRIAL: NCT01392040
Title: Clinical Validation of a New Algorithm for Computerized Dosing of Vitamin K Antagonist Therapy
Status: Completed | Type: Observational
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Alfonso Iorio, Dt, University Of Perugia
Other Study IDs: MIV_AI_10_001
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Anticoagulated Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients in oral anticoagulant therapy: Patients taking oral anticoagulant therapy

SUMMARY:
The purpose of this study is to determine whether the new algorithm is safety and effective in proposing the dosage and the timing of oral anticoagulant therapy.

ELIGIBILITY:
Inclusion Criteria:

* to take oral anticoagulant therapy for at least 2 years
* to be in stable conditions for at last 3 months

Exclusion Criteria:

* patients who need to perform surgery
* patients who interrupt therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the conditions for the patients inclusion are: to take oral anticoagulant therapy for at least 2 years; to be in stable conditions for at last 3 months
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-11; Primary Completion 2012-08 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Time spent in therapeutic range of INR by the patients | 6 months

SECONDARY OUTCOMES:
Thrombotic and bleeding events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michela Basileo, Dr, Principal Investigator — University Of Perugia; Alfonso Iorio, Dr, Principal Investigator — McMaster University
Locations (1):
- Hospital of Macerata, Macerata, Macerata, Italy